CLINICAL TRIAL: NCT01281293
Title: A Post Market, Long Term, Prospective, Observational, Multi-site Outcome Study to Follow the Clinical Course and Seizure Reduction of Patients With Refractory Seizures Who Are Being Treated With Adjunctive VNS Therapy.
Brief Title: Vagus Nerve Stimulation Clinical Outcomes Measured Prospectively in Patients Stimulated
Acronym: V-COMPAS
Status: Completed | Type: Observational
Sponsor: Cyberonics, Inc. (Industry)
Responsible Party: Sponsor
Organization: LivaNova (Industry)
Other Study IDs: Epilepsy (E)-103; E-103 (Other: Cyberonics)
Record Dates: First submitted 2011-01-05; First posted 2011-01-21 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Epilepsy
Keywords: V-COMPAS; Vagus Nerve Stimulation Clinical Outcomes;
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Vagus Nerve Stimulation (VNS) Therapy has been approved marked for the treatment of epilepsy since 1994. This post-market study is designed to follow the clinical course and outcomes for patients with refractory seizures treated with adjunctive VNS Therapy. Seizure frequency, seizure severity, side effects burden, depressive symptoms, global impressions, and health care utilization will be evaluated. The results of this study will provide data to guide physicians and their patients in the use of VNS Therapy for patients with refractory seizures who have failed initial trials of anti-epileptic drug (AED) therapy. The data being collected is not for the purposes of confirmatory assessment.

DETAILED DESCRIPTION:
Minimum ages eligible for the E-103 study is at least 7 years outside of the US, consistent with "Non-US" labeling and 12 years for sites in the US.

ELIGIBILITY:
Inclusion Criteria:

Patients enrolled in the study must meet all of the following criteria at Visit 1:

(Baseline) if Screening Incl/Excl is omitted:

1. Patients must agree to be treated with VNS Therapy. The decision to treat with VNS Therapy must have been made independent of and prior to participation in the study.
2. Patients participating at Sites not located in the US must follow the "Non-US" labeling and be at least 7 years or older and whose epileptic disorder is dominated by partial seizures (with or without secondary generalization) or generalized seizures that are refractory to antiepileptic medications; patients participating at Sites located in the United States must be 12 years or older and have partial onset seizures or must follow the indication for use statement (for VNS Therapy) in the country of origin.
3. Patient and/or caregiver must be able to give accurate seizure counts, health outcomes information, and complete study instruments with minimal assistance.
4. Patient or legal guardian understands study procedures and voluntarily signs an informed consent and in the United States a Health Insurance Portability and Accountability Act (HIPAA) authorization in accordance with institutional policies. In the event that the patient is under the age of 18 the patient will also be required to sign an assent affirming their agreement to participate in research according to local IRB requirements. Similar authorization is required per EC requirements, or equivalent authority.

   Additional Continuation Criteria to be evaluated at Visit 2 (Baseline):
5. Patient must be taking at least 1 anti-epileptic drug treatment and stable on said medications for at least 8 weeks (56 days) prior to baseline. (Rescue medication may be allowed on a case-by case basis with Cyberonics approval.)
6. Patient must have a minimum frequency of 3 seizures (excluding absence seizures, simple partial seizures and myoclonic jerks) per month (average over 2 months) prior to baseline; maximum frequency is 20 seizures per day.
7. Patient must have no more than 4 weeks between seizures (over 2 months) prior to baseline.

Exclusion Criteria:

Patients with any of the following will not be eligible for enrollment:

1. Patient currently uses, or is expected to use during the study, short-wave diathermy, microwave diathermy, or therapeutic ultrasound diathermy.
2. Patient is expected to require full body magnetic resonance imaging during the clinical study.
3. Patient has a progressive neurological condition (e.g. brain tumor etc.).
4. In the investigator's opinion, the inability of the patient, legal guardian or reluctance of the child to comply with the frequency of clinic visits during the treatment phase.
5. In the investigator's opinion, the patient has a history of noncompliance for seizure diary completion.
6. Patient is currently using an investigational device or pharmacologic medication not approved by either EU or US regulatory authority.
7. Patient has had a previous VNS Therapy implant.
8. In the investigator's opinion, the patient is suicidal.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of patients with a diagnosis of refractory seizures that are treated with adjunctive VNS Therapy.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2018-08-16 (Actual)

PRIMARY OUTCOMES:
Two-Year Clinical Follow-up | 27 months
  To follow the clinical course of patients with refractory seizures treated with adjunctive VNS Therapy over a two-year follow-up period.

SECONDARY OUTCOMES:
Efficacy and Safety | 27 months
  1. To evaluate over time the efficacy of best medical practice with adjunctive VNS Therapy in patients with refractory seizures.
  2. To evaluate over time the safety and tolerability of best medical practice with adjunctive VNS Therapy in patients with refractory seizures.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Jones, Study Director — LivaNova
Locations (20):
- United States (7):
  - Emory Healthcare, Atlanta, Georgia
  - University of Illinois College of Medicine at Peoria, Peoria, Illinois
  - University of Louisville Hospital, Louisville, Kentucky
  - Cornell University, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Covenant Hospital, Lubbock, Texas
  - St. Luke's Milwaukee, Milwaukee, Wisconsin
- UZ Gasthuisberg, Leuven, Belgium
- Germany (3):
  - Epilepsieklinik Tabor - Ladeburger Straße 15, Berlin
  - Albert-Ludwigs-Universität Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
- Sheba Medical Center, Ramat Gan, Israel
- United Kingdom (8):
  - Birmingham Children's Hospital, Birmingham
  - Foundation Trust Queen Elizabeth Hospital Birmingham, Birmingham
  - Southmead Hospital Bristol, Bristol
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - National Hospital for Neurology & Neurosurgery - UCLH, London
  - John Radcliffe Hospital, Oxford
  - Salford Royal Hospital, Salford
  - Royal Hallamshire Hospital, Sheffield